CLINICAL TRIAL: NCT05108922
Title: A Phase 3, Open-Label, Parallel-Group, 2-Arm Study to Investigate Amyloid Plaque Clearance With Donanemab Compared With Aducanumab-avwa in Participants With Early Symptomatic Alzheimer's Disease
Brief Title: A Study of Donanemab (LY3002813) Compared With Aducanumab in Participants With Early Symptomatic Alzheimer's Disease (TRAILBLAZER-ALZ 4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18369; I5T-MC-AACN (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer Disease
Keywords: Alzheimer's Disease with MCI or Mild Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — donanemab; aducanumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donanemab (Experimental): Donanemab is administered intravenously (IV) every 4 weeks (Q4W).
  Interventions: Drug: Donanemab
- Aducanumab (Active Comparator): Aducanumab administered IV per US label.
  Interventions: Drug: Aducanumab

INTERVENTIONS:
Drug: Donanemab — Participants received 700 milligram (mg) donanemab administered by intravenous (IV) infusion every 4 weeks (Q4W) for first three doses and then 1400 mg IV Q4W.
  Other Names: LY3002813
  Arms: Donanemab
Drug: Aducanumab — Participants received aducanumab administered by IV infusion per US label (prescribing information/routine clinical practice).
  Arms: Aducanumab

SUMMARY:
The main purpose of this study is to compare donanemab to aducanumab on brain amyloid plaque clearance in participants with early symptomatic Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in memory function reported by the participant or informant for ≥6 months.
* Meet florbetapir F18 PET scan criteria.
* A Clinical Dementia Rating (CDR)-Global Score of 0.5 or 1.
* Must consent to apolipoprotein E (ApoE) genotyping
* Must have a mini mental state examination (MMSE) score between 20 and 30
* Have a study partner who will provide written informed consent to participate, is in frequent contact with the participant (defined as at least 10 hours per week), and will accompany the participant to study visits or be available by telephone at designated times.
* Have adequate literacy, vision, and hearing for neuropsychological testing in the opinion of the investigator at the time of screening.
* Women not of childbearing potential may participate

Exclusion Criteria:

* Significant neurological disease affecting the central nervous system (other than AD), that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson's disease, multiple concussions, history of transient ischemic attack or stroke, or epilepsy or recurrent seizures (except febrile childhood seizures).
* Current serious or unstable medical illnesses including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, psychiatric (including actively suicidal or deemed at risk of suicide, or current alcohol or substance abuse), immunologic, infectious, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study; or has a life expectancy of approximately

  ≤24 months.
* History of clinically significant multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions (including but not limited to erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and/or exfoliative dermatitis).
* History of bleeding disorder or use of medications with platelet anti-aggregant or anti-coagulant properties (unless aspirin at ≤325 milligram (mg).
* Have had prior or current treatment with donanemab or aducanumab
* Have known allergies to donanemab or aducanumab, related compounds, or any components of the formulation
* Prior or current participation in any immunotherapy study targeting Amyloid beta

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-2559) or 1-317-615-4559 Mon - Fri 9 am - 5 pm Eastern time (UTC/GMT) - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- United States (31):
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Clinical Research, Irvine, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Charter Research - Lady Lake, Lady Lake, Florida
  - ClinCloud - Maitland, Maitland, Florida
  - ClinCloud - Viera, Melbourne, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Optimus U Corporation, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - Brain Matters Research, Stuart, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Columbus Memory Center, PC, Columbus, Georgia
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Donald S. Marks M.D., P.C., Plymouth, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Abington Neurological Associates, Ltd., Abington, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Kerwin Medical Center, Dallas, Texas
  - National Clinical Research, Inc, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Salloway S, Pain A, Lee E, Papka M, Ferguson MB, Wang H, Hu H, Lu M, Oru E, Ardayfio PA, Hoban DB, Collins EC, Brooks DA, Sims JR. TRAILBLAZER-ALZ 4: A phase 3 trial comparing donanemab with aducanumab on amyloid plaque clearance in early, symptomatic Alzheimer's disease. Alzheimers Dement. 2025 May;21(5):e70293. doi: 10.1002/alz.70293. PMID 40390253
- See also: A Study of Donanemab (LY3002813) Compared With Aducanumab in Participants With Early Symptomatic Alzheimer's Disease (TRAILBLAZER-ALZ 4) — https://trials.lillytrialguide.com/en-US/trial/7lW96VnHH5irho2IpKQCFM

RESULTS

PARTICIPANT FLOW:
Groups:
- Aducanumab: Participants received aducanumab administered by intravenous (IV) infusion per US label (prescribing information/routine clinical practice).
- Donanemab: Participants received 700 milligram (mg) donanemab administered by IV infusion every 4 weeks (Q4W) for first three doses and then 1400 mg IV Q4W.
Period: Overall Study
Arm/Group | Aducanumab | Donanemab
Started | 74 | 74
Received at Least One Dose of Study Drug | 69 | 71
Intermediate Tau Analysis Set | 28 | 27
Completed | 55 | 58
Not Completed | 19 | 16
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Inadvertent enrollment | 0 | 1
Not completed — Physician Decision | 2 | 3
Not completed — Protocol deviation | 1 | 0
Not completed — Screen failure | 1 | 0
Not completed — Withdrawal by Subject | 11 | 8

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Donanemab: Participants received 700 mg donanemab administered by IV infusion Q4W for first three doses and then 1400 mg IV Q4W.
- Total: Total of all reporting groups
Arm/Group | Aducanumab | Donanemab | Total
Number analyzed (Participants) | 69 | 71 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.70 (6.79) | 74.10 (6.87) | 73.40 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 27 | 33 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 65 | 67 | 132
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 61 | 71 | 132
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 71 | 140

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reach Complete Amyloid Plaque Clearance on Florbetapir F18 Positron Emission Tomography (PET) Scan (Superiority) on Donanemab Versus Aducanumab
Description: Amyloid deposition in the brain is one of the defining neuropathologic findings of Alzheimer's disease (AD). Amyloid PET scan assesses cerebral amyloid load using florbetapir tracer which is standardized into Centiloids for evaluation of AD. Florbetapir exhibits high affinity specific binding to amyloid plaques. Centiloid values on Centiloid scale is based on mean composite Standardized Uptake Value Ratio (SUVR) in cingulate, frontal, parietal and temporal cortexes using whole cerebellum as reference region. SUVR is ratio of tracer uptake in each of cingulate, frontal, parietal and temporal cortexes relative to cerebellum. Complete brain amyloid plaque clearance is a binary outcome and is defined as a Centiloid value <24.1 from the florbetapir F18 PET scan.
Time Frame: 6 Months
Population: All randomized participants who received at least one dose of study drug to donanemab or aducanumab with a baseline and at least one postbaseline Florbetapir F18 PET scan data at the primary outcome (6-month) database lock.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 64 | 66
Percentage of participants | 1.6 [0.0 to 4.6] | 37.9 [26.2 to 49.6]
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Analysis was based on logistic regression model with treatment, Apolipoprotein (ApoE) ε4 Carrier Status, baseline amyloid Level, baseline age as factors; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 29.26, 95% CI 2-sided [5.30 to 100.0]

2. Primary Outcome: Percentage of Participants Who Reach Complete Amyloid Plaque Clearance on Florbetapir F18 PET Scan in the Low/Medium (Intermediate) Subpopulation (Superiority) on Donanemab Versus Aducanumab
Description: Complete brain amyloid plaque clearance is a binary outcome and is defined as a Centiloid value <24.1 from the florbetapir F18 PET scan.
Time Frame: 6 Months
Population: All randomized participants who received at least one dose of study drug to donanemab or aducanumab with a baseline and at least one postbaseline Florbetapir F18 PET scan data and a baseline flortaucipir F18 PET scan meeting the low/medium tau criteria at the primary outcome (6-month) database lock.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 26 | 26
Percentage of participants | 3.8 [0.0 to 11.2] | 38.5 [19.8 to 57.2]
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Analysis was based on logistic regression model with treatment, ApoE ε4 Carrier Status, baseline amyloid Level, baseline age as factors; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 15.18, 95% CI 2-sided [2.04 to 100.0]

3. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) on Donanemab Versus Aducanumab
Description: Florbetapir PET imaging was used as a quantitative amyloid biomarker. Quantitative amyloid burden was first formalized as the average Standardized Uptake Value Ratio (SUVR) in six predetermined cortical areas of the brain relative to the cerebellum as a reference region. Larger SUVR reflects the larger cortical amyloid burden relative to cerebellum. SUVR values were further calibrated to a Centiloid (CL) scale. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. A negative change indicates an improvement from baseline.
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 64 | 66
Centiloids | -16.413 (3.7685) | -62.104 (3.6898)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, ANCOVA — Analysis between treatment group comparison p-value using analysis of covariance (ANCOVA) model for endpoint measures: Change (CHG) = Baseline + ApoE ε4 Carrier Status + Baseline Age + Treatment; LS Mean difference (Final Values) = -45.691, 95% CI 2-sided [-54.84 to -36.54], Standard Error of Mean 4.6132

4. Secondary Outcome: Mean Percent Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 6 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 64 | 66
Percent change | -16.956 (4.0253) | -65.169 (3.9412)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, ANCOVA — Analysis between treatment group comparison p-value using ANCOVA model for endpoint measures: Percent change (PCHG) = Baseline + ApoE ε4 Carrier Status + Baseline Age + Treatment; LS Mean difference (Final Values) = -48.213, 95% CI 2-sided [-57.99 to -38.44], Standard Error of Mean 4.9276

5. Secondary Outcome: Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan in the Low/Medium (Intermediate) Tau Subpopulation (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 26 | 26
Centiloids | -23.824 (7.7028) | -64.076 (7.3359)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, ANCOVA — Analysis between treatment group comparison p-value using ANCOVA model for endpoint measures: CHG = Baseline + ApoE ε4 Carrier Status + Baseline Age + Treatment; LS Mean difference (Final Values) = -40.252, 95% CI 2-sided [-61.87 to -18.64], Standard Error of Mean 10.5510

6. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 12 Months
Population: All randomized participants who received at least one dose of study drug to donanemab or aducanumab with a baseline and at least one postbaseline Florbetapir F18 PET scan data at the 12-month database lock.
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Centiloids | -56.06 (2.977) | -80.03 (2.973)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, Mixed Models Analysis — Analysis between treatment group comparison p-value using mixed model for repeated measures (MMRM) model for Treatment + Visit + Treatment*Visit + ApoE4 Carrier Status + Baseline Brain Amyloid Level + Baseline Age; LS Mean difference (Final Values) = -23.97, 95% CI 2-sided [-32.35 to -15.60], Standard Error of Mean 4.231

7. Secondary Outcome: Mean Percent Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 12 Months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Percent change | -56.97 (3.081) | -82.79 (3.077)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, Mixed Models Analysis — Analysis between treatment group comparison p-value using MMRM model for Treatment + Visit + Treatment*Visit + ApoE4 Carrier Status + Baseline Brain Amyloid Level + Baseline Age; LS Mean difference (Final Values) = -25.82, 95% CI 2-sided [-34.49 to -17.15], Standard Error of Mean 4.381

8. Secondary Outcome: Percentage of Participants Who Reach Complete Amyloid Plaque Clearance on Florbetapir F18 Positron Emission Tomography (PET) Scan (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 1
Time Frame: 12 Months
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Percentage of participants | 24.59 | 70.00
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, Regression, Logistic — Analysis was based on logistic regression model with 1 (Screening) value, ApoE4 Status, Age, Treatment, Time, and Treatment-by-time interaction as factors. Variance-Covariance structure = Unstructured; Odds Ratio (OR) = 8.38, 95% CI 2-sided [3.37 to 20.81]

9. Secondary Outcome: Percentage of Participants Who Reach Complete Amyloid Plaque Clearance on Florbetapir F18 PET Scan in the Low/Medium (Intermediate) Subpopulation (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 1
Time Frame: 12 Months
Population: All randomized participants who received at least one dose of study drug to donanemab or aducanumab with a baseline and at least one postbaseline Florbetapir F18 PET scan data and a baseline flortaucipir F18 PET scan meeting the low/medium tau criteria at the 12-month database lock.
Measure: Number; unit: percentage of participants
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 27 | 26
percentage of participants | 18.52 | 76.00
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < .001, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 37.73, 95% CI 2-sided [5.71 to 99.99]

10. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan in the Low/Medium (Intermediate) Tau Subpopulation (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 12 Months
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 27 | 26
Centiloids | -57.77 (4.419) | -84.53 (4.565)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = -26.75, 95% CI 2-sided [-39.78 to -13.73], Standard Error of Mean 6.479

11. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) on Donanemab 6 Months Versus Aducanumab 12 Months
Description: as for outcome 3
Time Frame: Baseline, 6 Months and 12 Months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Centiloids | -56.056 (2.9768) | -63.987 (2.8142)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p = 0.0558, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = -7.931, 95% CI 2-sided [-16.060 to 0.199], Standard Error of Mean 4.1187

12. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Non-inferiority) on Donanemab 6 Months Versus Aducanumab 12 Months
Description: as for outcome 3
Time Frame: Baseline, 6 Months and 12 Months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Centiloids | -56.056 (2.9768) | -63.987 (2.8142)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Non-Inferiority — Non-inferiority margin of interest: 5 Centiloids; Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = -7.931, 95% CI 2-sided [-16.060 to 0.199], Standard Error of Mean 4.1187

13. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 18 Months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Centiloids | -72.18 (2.883) | -84.22 (2.905)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = -12.04, 95% CI 2-sided [-20.19 to -3.88], Standard Error of Mean 4.120

14. Secondary Outcome: Time to Reach Complete Amyloid Plaque Clearance on Donanemab Versus Aducanumab
Description: Time to reach complete amyloid plaque clearance at 18 months was evaluated.
Time Frame: 18 Months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
days | 568.00 [542.00 to NA] — Upper limit of 95% confidence interval was not calculated as there were not enough events. | 359.00 [343.00 to 377.00]
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, Log Rank

15. Secondary Outcome: Mean Percent Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Superiority) Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 18 Months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
percent change | -72.84 (3.011) | -86.29 (3.030)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = -13.45, 95% CI 2-sided [-21.96 to -4.93], Standard Error of Mean 4.300

16. Secondary Outcome: Percentage of Participants Who Reach Complete Amyloid Plaque Clearance on Florbetapir F18 Positron Emission Tomography (PET) Scan (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 1
Time Frame: 18 Months
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
percentage of participants | 43.10 | 76.79
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 4.68, 95% CI 2-sided [1.93 to 11.34]

17. Secondary Outcome: Percentage of Participants Who Reach Complete Amyloid Plaque Clearance on Florbetapir F18 PET Scan in the Low/Medium (Intermediate) Subpopulation (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 2
Time Frame: 18 Months
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 27 | 26
percentage of participants | 43.48 | 72.00
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p = 0.022, Regression, Logistic — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 6.34, 95% CI 2-sided [1.32 to 30.54]

18. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan in the Low/Medium (Intermediate) Tau Subpopulation (Superiority) on Donanemab Versus Aducanumab
Description: as for outcome 3
Time Frame: Baseline, 18 Months
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 27 | 26
Centiloids | -72.24 (4.374) | -86.57 (4.408)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Superiority; p = 0.028, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = -14.33, 95% CI 2-sided [-27.07 to -1.59], Standard Error of Mean 6.333

19. Secondary Outcome: Mean Absolute Change From Baseline in Brain Amyloid Plaque on Florbetapir F18 PET Scan (Non-inferiority) on Donanemab 6 Months Versus Aducanumab 18 Months
Description: as for outcome 3
Time Frame: Baseline, 6 Months and 18 Months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Aducanumab | Donanemab
Number analyzed (Participants) | 65 | 67
Centiloids | -72.178 (2.8834) | -64.347 (2.8645)
Statistical Analysis 1: Comparison: Aducanumab vs Donanemab; Test type: Non-Inferiority — Non-inferiority margin of interest: 5 Centiloids; Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; LS Mean difference (Final Values) = 7.831, 95% CI 2-sided [-0.226 to 15.889], Standard Error of Mean 4.0870

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 76
Description: All randomized participants who received at least one dose of study drug to donanemab or aducanumab. Gender specific events only occurring in male or female participants have had the number of participants at Risk adjusted accordingly.
Arm/Group | Aducanumab | Donanemab
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/71
Serious Adverse Events (participants affected / at risk) | 8/69 | 13/71
Other Adverse Events (participants affected / at risk) | 59/69 | 58/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aducanumab (N=69) | Donanemab (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 2 (2) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Aducanumab (N=69) | Donanemab (N=71)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (3)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (4) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual field defect (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Parotid duct obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (3) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 3 (3) | 0 (0)
Infusion site reaction (General disorders) | 1 (1) | 3 (3)
Mass (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 13 (14) | 20 (22)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal foot infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (6) | 3 (3)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (5)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 7 (10)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Biopsy prostate (Investigations) | 0/27 (0) | 1/33 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0)
Vitamin b12 decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 17 (20) | 13 (14)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 23 (29) | 17 (21)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Brain fog (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 6 (9)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (11) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Superficial siderosis of central nervous system (Nervous system disorders) | 7 (7) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (3)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/27 (1) | 0/33 (0)
Testicular pain (Reproductive system and breast disorders) | 0/27 (0) | 1/33 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (6)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Epiretinal membrane peel (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 2 (3)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypertensive urgency (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 4 (5)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT05108922/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT05108922/SAP_001.pdf